CLINICAL TRIAL: NCT01371942
Title: Mutational Profiling in Colorectal Tumors to Determine Its Role in the Diagnosis, Prognostic Significance and Their Impact in Clinical Management
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Gi-Shih Lien, Department of Gastroenterology, Wanfang Hospital
Other Study IDs: 99064
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer(CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate mutational changes occurring in colorectal tumors, from benign polyps, malignant cancer and metastatic tumors. The investigators also plan to establish the clinical correlation, emphasizing on aspects such as the diagnosis and prognosis of disease and the specific treatment outcome. For the purpose, the investigators plan to obtain specimens from patients with colorectal tumors to extract DNA material. The specimens include tissues from either primary (mostly endoscopic biopsies specimens) or metastatic tumors (obtained from sonogram or other imaging modalities guided biopsy), as well as other humors including blood (for serum), malignant ascites, pleural effusions or other body fluids that could be related to CRCs. These patients would receive detailed explanations with regard to the investigations before signing IRB consent. At the initial stage, Wanfang Medical Center would be the only medical institution where endoscopic specimens would be collected. The project would eventually be extended to the Taipei Medical University Hospital and Shuan-Ho Hospital.

DETAILED DESCRIPTION:
The following are items corresponding to the critical tasks of the project.

1. Collect, annotate, and store fresh endoscopic specimens of suspicious abnormal tissue (premalignant lesions and primary tumors for genetic mutational investigation;
2. Collect, annotate, and store fresh specimens from metastatic lesions (e.g.: hepatic metastatic tumors), under sonographic or other imaging modalities guided biopsy procedures;
3. Collect, process, and store serum, plasma and isolate lymphocytes from blood drawn from patients with colorectal tumor;
4. Establish a database to link materials acquisition, pathologic, and clinical information on patients who participate in the protocol;
5. To utilize the clinical database to perform clinical and pathological correlation with the results of current and future scientific studies;
6. To evaluate genomic and biochemical alterations in colorectal tumors.
7. To test the effect of small molecule inhibitors on the activation of wild-type and mutant genetic alterations and/or other potential molecular targets.
8. To correlate tumor genotype and signaling abnormalities with clinical response to genetic alterations and/or other potential molecular targets inhibitors
9. Analysis of laboratory findings in relationship to patient demographics and clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been noted with a colonic tumor (benign polyps or colorectal cancer) on colonoscopy. Patients with lesions located other than the primary tumor (metastatic lesions) such as liver metastasis, enlarged lymph nodes suspicious of metastasis, malignant pleural effusion, ascites, etc. are also enrolled.
* Age 20
* Signed consent

Exclusion Criteria:

* Known HIV infection
* Known to have bleeding tendency, precluding for biopsy
* Any other clinical conditions, which, in the opinion of the principal investigator, would not allow completion of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-05; Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gi-Shih Lien, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan